CLINICAL TRIAL: NCT04982835
Title: M6-C Artificial Cervical Disc Two-Level IDE Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthofix Inc. (Industry)
Collaborators: Spinal Kinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-C003-Pivotal
Record Dates: First submitted 2019-09-17; First posted 2021-07-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervical Disc Degenerative Disorder
Keywords: artificial cervical disc; degenerative disc disease; total disc replacement; Spinal Kinetics
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Masking Description: Participants will be assigned a treatment group by enrolling site and will not be blinded to the treatment group assignment before their surgery. Investigator, and site will not be blinded to treatment assignment due to the need to prepare for the respective surgery associated with the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- M6-C Artificial Cervical Disc (Experimental): The M6-C is an investigational device composed of two outer and inner endplates made of titanium with a polycarbonate urethane nucleus (plastic center) and a polyethylene fiber annulus (strong thread-like binding). Around the polyethylene annulus is a polyurethane sheath (plastic cover). The outer endplates have keels to anchor the disc to bone. The outer endplates and keels are both coated with a titanium plasma spray. The M6-C is provided in two heights (6mm and 7mm) and four footprints (Medium, Medium Long, Large, Large Long).
  Interventions: Device: M6-C Artificial Cervical Disc
- Anterior Cervical Discectomy & Fusion (ACDF) (Active Comparator): ACDF will be performed using one of four FDA-approved anterior cervical plate systems and corticocancellous allograft bone. The four plating systems used in this study are:
  * Orthofix CETRA Anterior Cervical Plate System
  * Medtronic Sofamor/Danek Venture Anterior Cervical Plate System
  * DePuy Synthes: SKYLINE Anterior Cervical Plate System
  * Stryker Aviator Anterior Cervical Plating System
  Interventions: Device: ACDF

INTERVENTIONS:
Device: M6-C Artificial Cervical Disc — An incision will be made in the front of the neck and the damaged disc located between cervical vertebrae (neck bones) will be removed so that the M6-C artificial cervical disc can be placed into the space where the damaged disc was removed. This procedure will be performed using x-ray technology (fluoroscopy) guide the surgeon in placement of the M6-C in between the cervical vertebrae. This process will be repeated to replace the second damaged disc.
  Arms: M6-C Artificial Cervical Disc
Device: ACDF — One of four FDA-approved cervical plate systems will be used for the ACDF. An incision will be made in the front of the neck and the damaged disc located between cervical vertebrae (neck bones) will be removed. Then, a piece of donor bone will be placed in the space where the damaged disc was removed and a metal plate will be screwed into the bones above and below the disc. This procedure will be performed using x-ray technology (fluoroscopy) to guide the surgeon in the placement of the cervical plate system. This process will be repeated to treat the other damaged disc.
  Arms: Anterior Cervical Discectomy & Fusion (ACDF)

SUMMARY:
Prospective, concurrently controlled, multi-center study to evaluate the safety and effectiveness of the Spinal Kinetics M6-C™ artificial cervical disc compared to anterior cervical discectomy and fusion (ACDF) for the treatment of contiguous two-level symptomatic cervical radiculopathy at vertebral levels from C3 to C7 with or without spinal cord compression.

DETAILED DESCRIPTION:
Patients will be concurrently enrolled in the M6-C treatment group and the ACDF control group. Patients should have failed at least six weeks of conservative treatment or demonstrate progressive symptoms despite continued non-operative treatment. For the study, 263 patients will undergo either a two-level cervical artificial disc procedure, or an instrumented (ACDF) procedure as per site group assignment. Patients will be evaluated clinically, radiographically, and via the collection of patient-reported outcomes at 6 Weeks, 3 Months, 6 Months, 12 Months and 24 Months. The primary endpoint is Overall Success at 24 Months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of degenerative cervical radiculopathy with or without spinal cord compression requiring surgical treatment at two contiguous levels from C3 to C7 demonstrated by signs and/or symptoms of disc herniation and/or osteophyte formation (e.g. neck and/or arm pain, radiculopathy, etc.) and is confirmed by patient history and radiographic studies (e.g. MRI, CT, x-rays, etc.)
* Inadequate response to conservative medical care over a period of at least 6 weeks or have the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative management
* Neck Disability Index score of ≥ 30% (raw score of ≥ 15/50)
* Neck or arm pain Visual Analog Scale Score ≥ 4 on a scale of 0 to 10
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent
* Skeletally mature and at least 18 years old but not older than 75 years old

Exclusion Criteria:

* More than two cervical levels requiring surgery, or two non-contiguous levels requiring surgery
* Previous anterior cervical spine surgery
* Axial neck pain as the solitary symptom
* Previous posterior cervical spine surgery (such as a posterior element decompression) that destabilizes the cervical spine
* Advanced cervical anatomical deformity (such as ankylosing spondylitis, scoliosis) at either of the operative levels or adjacent levels
* Symptomatic facet arthrosis
* Less than four degrees of motion in flexion/extension at either of the index levels
* Instability as evidenced by subluxation greater than 3 millimeters at either of the index or adjacent levels as indicated on flexion/extension x-rays.
* Advanced degenerative changes (e.g., spondylosis) at either of the index vertebral levels as evidenced by bridging osteophytes, central disc height less than 4 millimeters and/or < 50% of the adjacent normal intervertebral disc, or kyphotic deformity > 11 degrees on neutral x-rays
* Severe cervical myelopathy (i.e., Nurick's Classification greater than 2)
* Active systemic infection or infection at the operative site
* Co-morbid medical conditions of the spine or upper extremities that may affect the cervical spine neurological and/or pain assessment
* Metabolic bone disease such as osteoporosis that contradicts spinal surgery
* History of an osteoporotic fracture of the spine, hip or wrist
* History of an endocrine or metabolic disorder (e.g. Paget's disease) known to affect bone and mineral metabolism
* Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
* Known allergy to titanium, stainless steels, polyurethane, polyethylene, or ethylene oxide residuals
* Fibromyalgia, Rheumatoid Arthritis (or other autoimmune disease), or a systemic disorder such as HIV or acute hepatitis B or C.
* Insulin dependent diabetes
* Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion
* Pregnant, or intend to become pregnant, during the course of the study
* Severe obesity (Body Mass Index greater than 45)
* Physical or mental condition (e.g. psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain or quality of life.
* Involved in current or pending spinal litigation where permanent disability benefits are being sought.
* Incarcerated at time of study enrollment
* Current participation in other investigational study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional Impairment - Neck Disability Index Score (NDI) | 24 Month
  Change in condition-specific functional impairment will be evaluated using a 10 item NDI outcomes questionnaire to assess change in the functional impairment score. NDI scores range from 0-50 (0%-100%) with higher scores demonstrating greater disability.
Overall Participant Success Rate (M6-C Artificial Cervical Disc) | 24 Month
  - Participant success is a composite endpoint of all of the listed Primary Outcome Measures.
- Serious Adverse Event(s) | 24 Month
  No serious adverse events classified as device or device procedure related (as determined by the Clinical Events Committee).
- Additional Surgical Intervention | 24 Month
  No supplemental surgical procedure at the index level(s) including supplemental fixation, revision and/or device removal.
- Neurologic Function | 24 Month
  Maintenance or improvement in neurological function as determined by Clinical Events Committee review of neurological exam results.

SECONDARY OUTCOMES:
Neck and Arm Pain | 24 Month
  Change in severity of neck and arm pain will be evaluated on a 10-cm Visual Analog Scale (VAS). Zero = no pain, 10 = worst possible pain.
Health-Related Quality of Life | 24 Month
  Maintenance or improvement of health-related quality of life will be evaluated using the SF-12v2 Health Survey.
Radiographic Assessments | 24 Month
  Quantitative and qualitative assessments compared to baseline evaluating surgical success outcomes for both cohorts.
FOSS Dysphagia Scale | 24 Month
  The five-stage Functional Outcome Swallowing Scale (FOSS) will be used to determine presence/absence of post-operative oropharyngeal dysphagia and severity of the disorder and outcome. On the 0 to 4 FOSS scale, 0=normal; asymptomatic, whereas 5=severe dysphagia; nonoral feeding.
Odom's Criteria | 24 Month
  Physician assessment of the clinical disposition of a participant at two-years using the 4-point rating scale (excellent, good, satisfactory, poor) for assessing the clinical outcome after cervical spine surgery.
Patient Satisfaction | 24 Month
  A brief Participant Satisfaction Questionnaire (very satisfied, satisfied, neutral, unsatisfied, very unsatisfied) regarding the outcome of their surgery at two-years.
Pain Medication Usage | 24 Months
  Change in usage of post-operative pain medications specifically prescribed for cervical spine will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Erturan, MD, JD, Study Director — Orthofix Inc.
Locations (21):
- United States (21):
  - Desert Institute for Spine Care, Phoenix, Arizona
  - Beverly Hills Spine Surgery, Beverly Hills, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Disc Sports & Spine Center, Newport Beach, California
  - UC Irvine Medical Center, Orange, California
  - Institute of Neuro Innovation, Santa Monica, California
  - St. Charles Spine Institute, Thousand Oaks, California
  - University of Colorado School of Medicine - Department of Orthopedics, Aurora, Colorado
  - Steadman Philipon Research Institute, Vail, Colorado
  - Orlando Health, Orlando, Florida
  - Joseph Spine Institute, Tampa, Florida
  - Longstreet Clinic, Gainesville, Georgia
  - Axis Spine, Coeur d'Alene, Idaho
  - Carle Health, Urbana, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Michigan Orthopedic Surgeons, Southfield, Michigan
  - The Orthopedic Center of St. Louis, St Louis, Missouri
  - Metropolitan Neurosurgery Associates - Englewood Health, Englewood, New Jersey
  - Mayfield Clinic, Cincinnati, Ohio
  - St. David's Healthcare, Austin, Texas
  - American Neurospine Institute/Medical City Frisco, Frisco, Texas

IPD SHARING:
Plan to Share IPD: No